CLINICAL TRIAL: NCT03852212
Title: Ninth Dorsal Osteopathic Visceral Manipulation D9 Affects Pancreas Blood Levels
Brief Title: Ninth Dorsal Osteopathic Visceral Manipulation D9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5548
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Osteopathia; Manipulation
Keywords: Thrust technique; Blood levels; Pancreas; Ninth vertebra; Manipulation
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group did not received any treatment
- Manipulation (Experimental): Experimental group received the osteopathic maneuver and the blood value were measured at baseline, after 2,5 and 10 minutes.
  Interventions: Other: Manipulation

INTERVENTIONS:
Other: Manipulation — Thrust technique application
  Arms: Manipulation

SUMMARY:
The aims of this study is to verify that the vertebral manipulation of dorsal level D9 influences the pancreas biochemical and endocrinology blood values.

DETAILED DESCRIPTION:
A longitudinal experimental study was conducted in which the osteopathic thrust maneuver was applied. In this research, 87 healthy subjects participated, of which 56.3% (n = 49) are men and 43.7% (n = 38) are women aged 19-29 who study at the Catholic University of Murcia.The blood analytical values of insulin and glycemia have been measured in 4 different times: at baseline, after 2,5 and 10 minutes of the technique application with the purpose to verify any possible change.

ELIGIBILITY:
Inclusion Criteria:

* students between 18-27 years old
* healthy persons
* Acceptance of informed consent

Exclusion Criteria:

* pancreatitis
* diabetes I,II type
* anemia
* Alcohol intake for 12 hours prior.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Basal insulin laboratory value change | 10 minutes
  The normal values of basal insulin measured with the imunoanalysis method are ˂ at 25.0 mU / l. If these values are exceeded, the effect of the manipulation in the study is verified
Basal glycemia laboratory value change | 10 minutes
  The normal values of basal glycemia measured with the enzymatic method vary between 60 - 105 mg / dl. The change of these values according to the reference laboratory has been the basis of the study.